CLINICAL TRIAL: NCT02859025
Title: Lateral Ramus Cortical Bone Plate in Alveolar Cleft Osteoplasty: Concomitant Use of Buccal Fat Pad Derived Cells and Autogenous Bone in a Preliminary Study
Brief Title: Concomitant Use of Buccal Fat Pad Derived Cells and Autogenous Bone in Alveolar Cleft Osteoplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arash Khojasteh, Associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sbmu9221
Record Dates: First submitted 2016-07-30; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Cleft of Alveolar Ridge
Keywords: Alveolar cleft; Osteoplasty; Tissue engineering; Stem cells; Regenerative medicine; Bone; Lateral ramus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A:Iiac (Active Comparator): Treated with anterior iliac crest spongy bone to fill defects, followed by coverage with collagen membrane.
  Interventions: Biological: anterior iliac crest graft
- B:MSCs+LRCP (Experimental): Treated with lateral ramus cortical bone plate (LRCP) to create a protected healing space by fixing it to adjacent walls of the cleft defect. BFPScs were loaded on NBBM and delivered to the defect
  Interventions: Biological: lateral ramus cortical bone+BFPSC+NBBM
- C:MSCs+liac (Experimental): Treated with anterior iliac crest spongy bone as in Group 1, but BFP-derived mesenchymal stem cells (MSCs ) cultured over NBBM were put over the spongy bone and covered with a collagen membrane.
  Interventions: Biological: anterior iliac crest graft+BFPSC+NBBM

INTERVENTIONS:
Biological: anterior iliac crest graft — Anterior iliac crest spongy bone filled the defects followed by coverage with collagen membrane.
  Arms: A:Iiac
Biological: lateral ramus cortical bone+BFPSC+NBBM — ramus cortical bone cage created a protected healing space and BFPSCs cultured over NBBM were put over the graft.
  Arms: B:MSCs+LRCP
Biological: anterior iliac crest graft+BFPSC+NBBM — Anterior iliac crest spongy bone filled the defects and BFPSCs cultured over NBBM were put over the spongy bone.
  Arms: C:MSCs+liac

SUMMARY:
Our aim was to combine regenerative techniques with bone grafting in human models to increase predictability and survival of reconstructed tissue. The MSCs in this study were derived from an intra oral fat source (BFP) and were cultured over natural bovine bone mineral granules and delivered within the lateral ramus cortical bone plate (LRCP)to treat human alveolar cleft defects.

DETAILED DESCRIPTION:
Patients enrolled in the present study were suffering from alveolar cleft and had previously received orthodontic treatment and only required secondary alveolar grafting. The buccal fat pad derived stem cells (BFPSCs) were harvested from buccal fat pad tissues of the patients. Patients were divided into 3 groups. Group A , the control group, was treated with anterior iliac crest (AIC) spongy bone to fill defects, followed by coverage with collagen membrane. Group B was treated with lateral ramus cortical bone cage (LRCP), used to create a protected healing space by fixing it to adjacent walls of the cleft defect. Group C was treated with (AIC) as in Group 1, but BFP-derived MSCs cultured over NBBM were put over the spongy bone and covered with a collagen membrane.Passage 3 BFPSCs were loaded on the implants ( Cerabone (Botiss, Berlin, Germany) a natural bovine bone mineral (NBBM); a granular biomaterial with a 200- to 850-µm particle size) 3 days prior to transplantation.Cone beam computed tomography (CBCT) was obtained after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral congenital cleft lip and palate
* Previous presurgical orthodontic treatment

Exclusion Criteria:

* History of malignancy
* History of radiation
* History of chemotherapy
* Pregnancy
* Systemic diseases contradicting dental and surgical treatments
* Conditions or drugs affecting bone remodeling or bone metabolism and connective tissue
* Allergy to collagen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
change in bone volume | before the surgery and 6 months after the surgery
  1-mm coronal sections of the treated region were taken before and after surgery, and new bone formation was assessed by CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentristry at Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Khojasteh A, Kheiri L, Behnia H, Tehranchi A, Nazeman P, Nadjmi N, Soleimani M. Lateral Ramus Cortical Bone Plate in Alveolar Cleft Osteoplasty with Concomitant Use of Buccal Fat Pad Derived Cells and Autogenous Bone: Phase I Clinical Trial. Biomed Res Int. 2017;2017:6560234. doi: 10.1155/2017/6560234. Epub 2017 Dec 12. PMID 29379800